CLINICAL TRIAL: NCT00871910
Title: A Phase 1 Dose-Escalation Study of the Safety, Pharmacokinetics, and Pharmacodynamics of the Cyclin-Dependent Kinase (CDK) Inhibitor SCH 727965 Administered Every 3 Weeks in Subjects With Advanced Malignancies
Brief Title: Phase 1 Every-3-Week Dosing of SCH 727965 in Patients With Advanced Cancer (Study P04630)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04630
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Solid Tumors; Lymphoma, Non-Hodgkin; Multiple Myeloma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Multiple Myeloma | interventions — dinaciclib; Aprepitant; Ondansetron; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 2 Hour SCH 727965 infusion (Experimental): Participants treated with 2 hour SCH 727965 IV infusion
  Interventions: Drug: SCH 727965
- 8 Hour SCH 727965 infusion (Experimental): Participants treated with 8 hour SCH 727965 IV infusion.
  Interventions: Drug: SCH 727965
- 24 Hour SCH 727965 infusion (Experimental): Participants treated with 24 hour SCH 727965 IV infusion.
  Interventions: Drug: SCH 727965
- 2 Hour SCH 727965 infusions plus aprepitant in Cycle 1 (Experimental): Participants randomized to 2 Hour SCH 727965 infusion, plus concomitant ondansetron and dexamethasone in Cycles 1 and 2, and aprepitant in Cycle 1 only.
  Interventions: Drug: SCH 727965; Drug: Aprepitant; Drug: Ondansetron; Drug: Dexamethasone
- 2 Hour SCH 727965 infusion plus aprepitant in Cycle 2 (Experimental): Participants randomized to 2 Hour SCH 727965 infusion, plus concomitant ondansetron and dexamethasone in Cycles 1 and 2, and aprepitant in Cycle 2 only.
  Interventions: Drug: SCH 727965; Drug: Aprepitant; Drug: Ondansetron; Drug: Dexamethasone

INTERVENTIONS:
Drug: SCH 727965 — SCH 727965 2 hour IV infusion on Day 1 of each 3 week cycle, administered in dose-escalating cohorts (Part 1 of the trial)
  Arms: 2 Hour SCH 727965 infusion
Drug: SCH 727965 — SCH 727965 8 hour IV infusion on Day 1 of each 3 week cycle,in dose-escalating cohorts
  Arms: 8 Hour SCH 727965 infusion
Drug: SCH 727965 — SCH 727965 24 hour IV infusion on Day 1 of each 3 week cycle, in dose-escalating cohorts
  Arms: 24 Hour SCH 727965 infusion
Drug: SCH 727965 — SCH 727965 29.6 mg/m2 2 hour IV infusion on Day 1 of each 3 week cycle
  Arms: 2 Hour SCH 727965 infusion plus aprepitant in Cycle 2; 2 Hour SCH 727965 infusions plus aprepitant in Cycle 1
Drug: Aprepitant — Oral aprepitant in Cycle 1 or Cycle 2, depending on the study arm: 125 mg 1 hour prior to the SCH 727965 infusion on Day 1, and 80 mg on Days 2 and 3.
  Other Names: Emend
  Arms: 2 Hour SCH 727965 infusion plus aprepitant in Cycle 2; 2 Hour SCH 727965 infusions plus aprepitant in Cycle 1
Drug: Ondansetron — Ondansetron 32 mg IV 30 minutes prior to the SCH 727965 infusion on Day 1 of Cycles 1 and 2.
  Other Names: Zofran
  Arms: 2 Hour SCH 727965 infusion plus aprepitant in Cycle 2; 2 Hour SCH 727965 infusions plus aprepitant in Cycle 1
Drug: Dexamethasone — Oral dexamethasone in Cycles 1 and 2: 12 mg 30 minutes prior to the SCH 727965 infusion on Day 1, and 8 mg in the morning on Days 2, 3, and 4.
  Other Names: Decadron
  Arms: 2 Hour SCH 727965 infusion plus aprepitant in Cycle 2; 2 Hour SCH 727965 infusions plus aprepitant in Cycle 1

SUMMARY:
Part 1 and Part 2 of this trial will evaluate the safety, tolerability, maximum administered dose, and dose limiting toxicity of SCH 727965 administered every 3 weeks as a 2 hour intravenous (IV) infusion (Part 1), and as an 8-hour or 24-hour IV infusion (Part 2). Each 3-week period is considered one treatment cycle. Part 3 of this trial will evaluate the effect of coadministration of antiemetic drug aprepitant on the pharmacokinetics of SCH 727965 administered as a 2 hour IV infusion once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, either sex, any race.
* Subjects must have histologically proven solid tumors, non-Hodgkin's lymphoma, or multiple myeloma.
* There must be no known standard therapy, or disease must be refractory to standard therapy.
* Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
* Adequate hematologic, renal, and hepatic organ function and laboratory parameters.

Exclusion Criteria:

* Symptomatic brain metastases or primary central nervous system malignancy.
* Previous radiation therapy to >25% of the total bone marrow.
* Previous treatment with SCH 727965.
* Known HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-10-11 (Actual); Primary Completion 2010-02-22 (Actual); Study Completion 2010-02-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SCH 727965, including maximum administered dose and dose-limiting toxicity | End of trial
In Part 1 and Part 2, pharmacodynamic effects of SCH 727965 with an ex vivo lymphocyte stimulation assay of participant's peripheral blood lymphocytes. | Cycle 1

SECONDARY OUTCOMES:
In Part 3, area under the plasma concentration versus time curve and maximum concentration of SCH 727965 administered as a 2 hour intravenous infusion with or without aprepitant in participants with advanced malignancies. | Cycle 1 Days 1 and 2, and Cycle 2 Days 1 and 2

REFERENCES:
- [Result] Zhang D, Mita M, Shapiro GI, Poon J, Small K, Tzontcheva A, Kantesaria B, Zhu Y, Bannerji R, Statkevich P. Effect of aprepitant on the pharmacokinetics of the cyclin-dependent kinase inhibitor dinaciclib in patients with advanced malignancies. Cancer Chemother Pharmacol. 2012 Dec;70(6):891-8. doi: 10.1007/s00280-012-1967-y. Epub 2012 Oct 9. PMID 23053255
- [Result] Mita MM, Mita AC, Moseley JL, Poon J, Small KA, Jou YM, Kirschmeier P, Zhang D, Zhu Y, Statkevich P, Sankhala KK, Sarantopoulos J, Cleary JM, Chirieac LR, Rodig SJ, Bannerji R, Shapiro GI. Phase 1 safety, pharmacokinetic and pharmacodynamic study of the cyclin-dependent kinase inhibitor dinaciclib administered every three weeks in patients with advanced malignancies. Br J Cancer. 2017 Oct 24;117(9):1258-1268. doi: 10.1038/bjc.2017.288. Epub 2017 Aug 31. PMID 28859059